CLINICAL TRIAL: NCT05749328
Title: Effect of Preoperative Oral Carbohydrate Shortening the Fasting Period on Hypotension After Anesthesia Induction in Elderly Patients With Joint Replacement
Brief Title: Effect of Preoperative Oral Carbohydrate on Hypotension After Anesthesia Induction in Elderly Patients With Joint Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022-0949
Record Dates: First submitted 2022-12-15; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-12

CONDITIONS: Carbohydrates; Aged; Post-induction Hypotension
MeSH Terms: interventions — Carbohydrates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbohydrate group (Experimental): Fasting at 20:00 on the eve of surgery, give 800ml of carbohydrate drink, the patient drinks freely, no more than 200ml per hour, to 3h before surgery, give carbohydrate drink again, according to 5ml/kg calculated dose, maximum 400ml, drink within 30 minutes.
  Interventions: Dietary Supplement: Carbohydrate
- Contral group (No Intervention): Fasting at 20:00 on the eve of surgery, fasting at 24:00, until the induction of anesthesia on the day of surgery

INTERVENTIONS:
Dietary Supplement: Carbohydrate — To ensure the safety of the trial, preoperative gastric ultrasound measurements will be performed on all patients to assess their gastric volume. See above for other details
  Arms: Carbohydrate group

SUMMARY:
The goal of this Randomized controlled trial is to investigate the effect of shortening the duration of preoperative oral carbohydrate drinks on blood pressure after anesthesia induction in elderly patients undergoing joint replacement surgery. The main question it aims to answer is Whether preoperative oral carbohydrate drinks can reduce the incidence of hypotension after anesthesia-induced hypotension in elderly patients undergoing joint replacement surgery.According to the numerical table method, the patients in the experimental group will drink carbohydrate drinks the night before the operation and 3 hours before the operation, and the control group patients will routinely fast

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective unilateral joint replacement (total hip or knee)
2. ASAⅠ-Ⅲ

Exclusion Criteria:

1. Diagnosed patients at high risk of reflux aspiration (diabetes mellitus, obesity (BMI>30), gastrointestinal obstruction, elevated intracranial pressure, and esophageal disease)
2. Eating disorders
3. History of gastrointestinal or epigastric surgery
4. Recent use of drugs that affect gastrointestinal motility
5. Heart disease (severe arrhythmias, severe heart valve disease, heart failure, unstable angina on the day of surgery)
6. Severe poorly controlled hypertension (MAP≥135 mmHg) or hypotension (MAP≤55 mmHg) before induction
7. Difficult airway
8. Severe hepatic and renal insufficiency

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypotension | 20 minutes after induction of anesthesia
  No surgical manipulation is performed within 20 minutes

SECONDARY OUTCOMES:
Duration of fasting and drinking | 1 day before the operation
Antral cross-sectional area | 30 minutes before anesthesia induction
Incidence of hypotension | during the whole operation
The dosage of vasoactive drugs | 20 minutes after induction of anesthesia
Thirst and hunger VAS score | 3 hours before and 1 day after the operation
Fasting blood glucose and insulin resistance index | 3 hours before the operation
Incidence of nausea and vomiting | 1 day after the operation

CONTACTS AND LOCATIONS:
Overall Officials: min yan, prof., Study Chair — The second affiliated hospital of Zhejiang University hangzhou

IPD SHARING:
Plan to Share IPD: No